CLINICAL TRIAL: NCT06357078
Title: The Effect of Art Therapy in Reducing Stress and Anxiety of Caregivers
Brief Title: Art Therapy and Caregivers Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amasya University (Other)
Responsible Party: Principal Investigator, Neşe Uysal, Principal Investigator, Amasya University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AmasyaU-NU-679
Record Dates: First submitted 2024-04-04; First posted 2024-04-10 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-04

CONDITIONS: Caregiver Stress Syndrome
MeSH Terms: interventions — Art Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Art Therapy (Experimental): Caregivers in the art therapy group will be given art therapy practices, lasting approximately 45 minutes-1 hour, twice a week for 4 weeks. Visual and handicraft practices (painting work, collage work, mandala work, painting with felt, clay work, painting and storytelling) are done in art therapy activities that will last for 4 weeks, and it is aimed to develop personal and emotional awareness, reduce stress and increase general well-being.
  Interventions: Other: Art Therapy
- Control (No Intervention): No intervention will be applied to the patients in the control group during the follow-up period, only data collection forms will be applied.

INTERVENTIONS:
Other: Art Therapy — Caregivers in the art therapy group will be given art therapy practices, lasting approximately 45 minutes-1 hour, twice a week for 4 weeks. Visual and handicraft practices (painting work, collage work, mandala work, painting with felt, clay work, painting and storytelling) are done in art therapy activities that will last for 4 weeks, and it is aimed to develop personal and emotional awareness, reduce stress and increase general well-being.
  Arms: Art Therapy

SUMMARY:
This research will be conducted to determine the effect of art therapy on the stress, anxiety and well-being of caregivers in the palliative care service.

DETAILED DESCRIPTION:
Introduction and aim: Evidence for the use of art in health promotion has been increasing in recent years. However, in the literature review, no study was found in our country examining the effect of art therapy on caregivers. In palliative care, the management of psychological problems such as stress and anxiety that caregivers frequently experience is very important for the health and quality of life of both the patient and the caregiver. Accordingly, this research will be conducted to determine the effect of art therapy on the stress, anxiety and well-being of caregivers in the palliative care service.

Methods: The research will be carried out as a randomized controlled experimental study in the palliative care unit of a training and research hospital. A distress thermometer will be applied to individuals who are primary caregivers of patients hospitalized in the palliative care unit, and caregivers with a stress score of 4 and above will be included in the sample. The block randomization method will be used in assigning the individuals included in the sample to the art therapy and control groups. Caregivers in the art therapy group will be given art therapy practices, lasting approximately 45 minutes-1 hour, twice a week for 4 weeks. Visual and handicraft practices (painting work, collage work, mandala work, painting with felt, clay work, painting and storytelling) are done in art therapy activities that will last for 4 weeks, and it is aimed to develop personal and emotional awareness, reduce stress and increase general well-being. Research data will be collected using Descriptive Information Form, Distress Thermometer, State Anxiety Inventory and Personal Well-Being Scale.

Conclusions: It is thought that this study will increase attention to art therapy, improve stress and anxiety levels in caregivers, and strengthen current and future research in art therapy and nursing research. Given the key role caregivers play in palliative care, it is important to support caregivers as a necessity for holistic and comprehensive health care services

ELIGIBILITY:
Inclusion Criteria:

* The age of 18 and over,
* Must be able to read and speak Turkish
* Care givers of patients hospitalized in palliative care clinics,
* Has a distress score of 4 or above,
* Does not have any sensory or cognitive health problems that would prevent communication,
* Must agree to participate in the study

Exclusion Criteria:

* No primary caregiver role
* Has a physical disability to perform artistic practices,

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2024-01-02 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Distress Thermometer | 4 weeks
  Distress Thermometer: Distress Thermometer is a Likert-type scale with scores from 0 (no stress) to 10 (extreme stress) and was developed to determine psychological distress. With the scale, which is short and easy to understand, individuals can easily mark their own stress levels within the ranges specified on the thermometer. The recommended cut-off point for the stress thermometer is 4 and above, and a score of 4 and above indicates the presence of stress.
The State Anxiety Inventory | 4 weeks
  The State Anxiety Inventory is a tool that is sensitive to affective, physiological and cognitive processes such as anxiety, anxiety and excitement, and is very sensitive to sudden changing reactions. There are reverse coded expressions in the scale (items 1, 2, 5, 8, 10, 11, 15, 16, 19 and 20). In evaluating the scale scores, after finding the separate total weights of the direct and reverse expressions, the total weight score of the reverse expressions is subtracted from the total weight score obtained for the direct expressions, and a predetermined, unchanging value is added to this number. The last value obtained is the individual's anxiety score. The total score obtained from the scale varies between 20-80, a high score indicates a high level of anxiety, and a low score indicates a low level of anxiety
Personal Well-Being Index | 4 weeks
  Personal Well-Being Index is a scale that measures happiness and well-being in individuals' lives. It is a thematic and 11-point Likert type (0: I am completely dissatisfied-5: I am neutral-10: I am completely satisfied) measurement tool that aims to measure individuals' satisfaction levels with eight living areas. The eight life domains are listed as personal health, success in life, personal relationships, personal security, social bond/belonging, standard of living, future certainty, and spirituality/religion. The scale includes a single question for each of the eight life domains. The lowest score that can be obtained from the scale is 0 and the highest score is 80. A high score from the scale indicates a high perception of personal well-being

CONTACTS AND LOCATIONS:
Locations (1):
- Neşe Uysal, Amasya, Turkey (Türkiye)